CLINICAL TRIAL: NCT05546606
Title: CO2 Removal in Severe Acute exacerbatIons of Chronic Obstructive Lung Diseases
Acronym: CORAIL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government); Xenios AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P150913J; 2022-A01343-40 (Other: Agence Nationale de sécurité du médicament et des produits de santé); PHRC-15-557 (Other Grant/Funding Number: French ministry of health)
Record Dates: First submitted 2022-09-15; First posted 2022-09-21 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-06

CONDITIONS: COPD Acute Exacerbation
Keywords: ECCO2R; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Prospective, multi-centre, randomized, controlled, open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single standard of care (No Intervention): COPD patients who require respiratory support for severe acute exacerbation (AE), either with NIV or with IMV.
- Strengthen standard of care reinforced with ECCO2R (Other): COPD patients who require respiratory support for severe acute exacerbations (AE), either with NIV or with IMV reinforced with ECCO2R
  Interventions: Device: ECCO2R

INTERVENTIONS:
Device: ECCO2R — ECCO2R therapy using the Xenios platform, CE-marked medical device of the firm Xenios AG (Heilbronn, Germany), including the following components: Xenios console, iLA active iLA Kit IPS and Novaport Twin (18Fr, 22Fr or 24 Fr) cannulas The maximal duration of ECCO2R therapy with one circuit will be of 29 days in agreement with the regulatory approval of the patient kit.
  Arms: Strengthen standard of care reinforced with ECCO2R

SUMMARY:
The aim of the study is to determine which standard of care strategy will best benefit very severe Acute Exacerbation (AE) of Chronic Obstructive Pulmonary Disease (COPD), single versus reinforced with ECCO2R and assess the respective efficacy and the safety. Very severe AE of COPD will be defined by high risk of Non-Invasive Ventilation (NIV) failure defined by need of intubation and/or in-Intensive Care Unit (ICU) mortality (Stratum 1) or by Invasive Mechanical Ventilation (IMV) after NIV failure and/or with severe hyperinflation and hypercapnia (Stratum 2).

DETAILED DESCRIPTION:
After inclusions, all patients from Stratum 1 (at high risk of NIV failure) and Stratum 2 (Intubation-IMV) will be randomly assigned to the single standard of care treatment or to the strengthen standard treatment reinforced with ECCO2R . Weaning of IMV in the strengthen standard of care group will precede weaning of ECCO2R. Weaning of NIV in the strengthen standard of care group will precede weaning of ECCO2R, except for patients with long-term NIV. The patients will undergo a maximum of 33 visits over the 1-year study duration, split in 3 successive periods: selection period, treatment period (until the discharge of the ICU or day 28 after randomisation), follow-up period after the discharge of the ICU (or after day 28) up to 1 year (after randomisation).

Selection period: before randomisation, demographics, medical and surgical history, clinical examination (including physical examination, respiration rate, encephalopathy score, sedation score, pain assessment, Simplified Acute Physiology Score 2, central body temperature, systolic and diastolic blood pressures, heart rate), blood sampling, electrocardiogram and ventilator parameters will be recorded.

Follow-up period: ECCO2R will start as soon as possible after randomisation in patients allocated to the strengthen standard of care group. All patients will be evaluated 12 + 2 hours after randomisation, followed by a daily visit with the collection of the following data if applicable: clinical examination, ECCO2R parameters, ventilator parameters, concomitant medications (including sedative drugs), occurrence of adverse events, date, time and criteria if endotracheal intubation (stratum 1). Arterial blood gases, hematology and serum biochemistry parameters will be assayed daily.

End of Research period: all patients will be evaluated at day 60 (+ 7 days), Day 90 (+ 7 days), Day 180 (+ 7 days) and 1 year (+ 7 days) at least by phone contact, with collection of: vital status, functional status (Severely Disabled or not, Katz Index of Independence in Activities of Daily Living), date of ICU discharge (if > Day 28), date of hospital discharge, occurrences of ICU re-admissions, of adverse events, type and length of mechanical ventilation needed if applicable.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Known or suspected diagnosis of COPD based on clinical history, pulmonary function test when available, arterial blood gases, physical examination, and chest radiograph
* Worsening dyspnea for < 2 weeks
* Written informed consent signed by patients or their surrogates, with possibility of an emergency procedure with deferred consent
* Patient affiliated to a Social Security System (excluding "AME: aide médicale d'état")
* Negative serum or urinary β-hCG for women of child-bearing potential
* Very severe AE criteria defined either by:

  1. Stratum 1: high likelihood of NIV failure defined by PaCO2 > 55 mmHg and pH < 7.25, either at baseline and/or after at least one hour of NIV
  2. Stratum 2: intubation and IMV since less than 72 hrs, either after NIV failure and/or with pH < 7.30 and PaCO2 > 55 mmHg and PEEPi (end-expiratory occlusion) > 5 cmH2O, while on Assist-Controlled Ventilation with the following parameters: VT: 8 ml/kg, RR: 12/min., applied PEEP: 0 cmH2O

Exclusion Criteria:

* Hemodynamic instability
* Known allergy to heparin or to any of the excipients of the specialty used
* Contra-indications to heparin listed in the SmPC of the specialty used.
* History of type II Heparin-induced thrombocytopenia
* Thrombocytopenia (platelets < 100.000/mm3)
* Recent major surgery
* Haemorrhagic disorders such as:

  * Organic lesion likely to bleed
  * Bleeding manifestations or tendencies linked to disorders of hemostasis
  * Intracerebral hemorrhage
* Uncontrolled arrhythmia
* Bleeding diathesis
* Body Mass Index > 35 kg/m2
* PaO2/FiO2 < 180 mmHg
* Do not intubate order
* Fibrosing idiopathic interstitial pneumonitis (based on the available medical files)
* Neuromuscular diseases (based on the available medical files)
* Patients with tracheotomy
* Patients with severe concomitant chronic systemic disease with a limited probability of survival (< 6 months)
* Severely disabled (confinement to bed and inability to wash or dress alone) patients before AE
* Pregnant woman
* Participation in another interventional study involving human participants up to their ICU discharge, whether the studies include an investigational medical device, or being in the exclusion period at the end of a previous study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-04-18 (Actual); Primary Completion 2024-05-11 (Actual); Study Completion 2025-03-11 (Estimated)

PRIMARY OUTCOMES:
Mortality rate | Up to 60 days
  To determine the best strategy between strengthen standard of care reinforced with ECCO2R, versus single standard of care,

SECONDARY OUTCOMES:
Invasive Ventilator-free days (IVFDs) | at 28 and 60 days
  To assess the efficacy of ECCO2R, based on the time on IMV
Ventilator-free days (VFDs), including both IVFDs and non-invasive ventilator-free days (NIV-VFDs) | at 28 and 60 days
  To assess the efficacy of ECCO2R, based on the time on IMV
28 day, 90 day, 180 day and 1 year all-cause mortality rate | Up to 1 year
  To assess the efficacy of ECCO2R, based on the all-cause mortality
Length of ECCO2R therapy | Up to 28 days
  To assess the efficacy of ECCO2R, based on ECCO2R device's performance
Proportion of patients without intubation and IMV (intubation and IMV avoided) | Up to 28 days
  To assess the efficacy of ECCO2R, based on intubation rate
Number of days with active mobilization (outside the bed) | Up to 28 days
  To assess the efficacy of ECCO2R, based on the ability to actively mobilize the patients
Rate of inability to wean from IMV | at Day 28 and Day 60
  To assess the safety, based on central venous catheter-related complications
Rate of ventilator associated pneumonia | at Day 28 and Day 60
  To assess the safety, based on central venous catheter-related complications
Rate of central venous catheter infection | Up to 28 days
  To assess the safety, based on ECCO2R-related complications,
Rate of deep venous thrombosis | Up to 28 days
  To assess the safety, based on ECCO2R-related complications,
Rate of vascular injury caused by cannulation | Up to 28 days
  To assess the safety, based on ECCO2R-related complications,
Rate of severe bleeding (any cause) | Up to 28 days
  To assess the safety, based on ECCO2R-related complications,
Rate of severe hemolysis | Up to 28 days
  To assess the safety, based on ECCO2R-related complications,
Rate of heparin-induced thrombocytopenia - type II | Up to 28 days
  To assess the safety, based on ECCO2R-related complications,

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc MD Diehl, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (20):
- France (20):
  - CHU Angers, Angers
  - CHU Besançon, Besançon
  - Hôpital Avicennes, AP-HP, Bobigny
  - CHD de Vendée, La Roche-sur-Yon
  - CH Le Mans, Le Mans
  - Hôpital de la Croix-Rousse, Lyon
  - Hôpital Nord, Marseille
  - CHU Lapeyronie, Montpellier
  - CHR Orléans, Orléans
  - Hôpital La Pitié Salpêtrière, AP-HP, Paris
  - Hôpital Cochin - APHP, Paris
  - Hôpital européen Georges Pompidou - APHP, Paris
  - Hôpital Tenon, Paris
  - CHU la Milétrie, Poitiers
  - CHU Pontchaillou, Rennes
  - CHU Rouen, Rouen
  - Centre Hospitalier de Saint Denis, Saint-Denis
  - Nouvel Hôpital Civil Strasbourg, Strasbourg
  - CHRU Bretonneau, Tours
  - Hôpital d'Instruction des Armées Robert Picqué, Villenave-d'Ornon

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol, ICF
Time Frame: One year after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on scientific project and scientific involvement of the PI team. The founder could be involved in the decision.
  Teams wishing obtain IPD must meet the sponsor and IP team to present scientifics (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractualization.